CLINICAL TRIAL: NCT00598013
Title: A Randomized Controlled Trial of Pioglitazone on Insulin Resistance, Insulin Secretion and Atherosclerosis in Renal Allograft Recipients Without History of Diabetes
Brief Title: Effect of Pioglitazone on Insulin Resistance and Atherosclerosis in Renal Allograft Recipients Without Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hyun Chul Lee, Professor, Department of internal medicine, Yonsei University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2004-0082; 82-2-2228-1930
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Kidney Transplantation; Insulin Resistance; Atherosclerosis
Keywords: Kidney Transplantation; Thiazolidinediones; Insulin Resistance; Atherosclerosis
MeSH Terms: conditions — Insulin Resistance; Atherosclerosis | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pioglitazone
- 2 (No Intervention)

INTERVENTIONS:
Drug: Pioglitazone — The pioglitazone treatment group received 30mg pioglitazone at 2 weeks after renal transplantation for 12 months.
  Arms: 1

SUMMARY:
The aim of this study was to evaluate the effect of pioglitazone treatment on insulin secretion, insulin resistance, and progression of atherosclerosis in renal allograft recipients without preoperative history of diabetes.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label study. The pioglitazone treatment group received 30mg pioglitazone at 2 weeks after renal transplantation for 12 months.

After treatment, we estimated insulin sensitivity index for transplantation,first phase and second phase insulin secretion, secretion area under the curve,and carotid intima-media thickness.

ELIGIBILITY:
Inclusion Criteria:

* Renal allograft recipients were eligible to participate in the study if they were aged ≥ 18 years, had no previous history of organ transplantation and were not currently using steroids or other immunosuppressants.

Exclusion Criteria:

* Diabetes before transplantation
* Severe metabolic or infectious disease
* Hepatic disease
* Congestive heart failure (New York Heart Association II-IV)
* Cadaver donor kidney donor transplantation
* Unstable condition of the transplanted kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2004-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance and Insulin Secretion | 1 year

SECONDARY OUTCOMES:
carotid intima-media thickness | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Chul Lee, Doctor, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882
- [Derived] Han SJ, Hur KY, Kim YS, Kang ES, Kim SI, Kim MS, Kwak JY, Kim DJ, Choi SH, Cha BS, Lee HC. Effects of pioglitazone on subclinical atherosclerosis and insulin resistance in nondiabetic renal allograft recipients. Nephrol Dial Transplant. 2010 Mar;25(3):976-84. doi: 10.1093/ndt/gfp567. Epub 2009 Oct 28. PMID 19875376